CLINICAL TRIAL: NCT02993354
Title: Noninvasive Monitoring of Uterine Electrical Activity and Fetal Heart Rate: A New External Monitoring Device
Acronym: EUM
Status: Completed | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-4881
Record Dates: First submitted 2016-12-12; First posted 2016-12-15 (Estimated); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Contraction

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Pregnant women: Pregnant women with singleton pregnancy with gestational age greater than or equal to 24 weeks.
  Interventions: Device: The EUM300 (electrical uterine myography)

INTERVENTIONS:
Device: The EUM300 (electrical uterine myography) — This study involves monitoring one group of pregnant women for contractions simultaneously using two different devices to determine if one is superior: the usual tocodynamometer commonly used. Women are simultaneously monitored with both devices.

SUMMARY:
The EUM (electrical uterine myography) (OB Tools, Israel) was tested and found to be reliable as a non-invasive method for evaluating uterine contractions and the fetal heart rate. It is safe and effective in monitoring uterine contractions. The investigators propose to perform a study to validate the accuracy and clinical usefulness of the EUM device by simultaneously monitoring obese patients with current method of external tocodynamometry with the EUM device. Providers will be blinded to the results of the EUM device. Caregivers will continue care as per current guidelines using the information obtained from the current monitoring methods. Information obtained from the EUM devices will not be used to determine the clinical course of action.

DETAILED DESCRIPTION:
Purpose:

The investigators propose to perform a study to validate the accuracy and clinical usefulness of the EUM device by comparing it with simultaneous use of current methods (external tocodynamometry) among obese patients.

Objective:

Compare the interpretability of the contractions recorded using the EUM device vs. those obtained from external tocodynamometer among obese pregnant women.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age >18 years old
2. Singleton pregnancy
3. Gestational age of 24 completed weeks or greater based on the estimated due date as calculated from last menstrual period or early ultrasound
4. Category I (reassuring) fetal heart rate tracing at time of enrollment

Exclusion Criteria:

1. Fetal anomaly or chromosome defect
2. Allergy to silver
3. Woman with implanted electronic device of any kind
4. Irritated skin or open wound on the abdominal wall

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant women
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2021-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bernstein, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Jack D. Weiler Hospital of Montefiore Medical Center, The Bronx, New York, United States

REFERENCES:
- [Derived] Moni SS, Kirshenbaum R, Comfort L, Kuba K, Wolfe D, Xie X, Negassa A, Bernstein PS. Noninvasive monitoring of uterine electrical activity among patients with obesity: a new external monitoring device. Am J Obstet Gynecol MFM. 2021 Jul;3(4):100375. doi: 10.1016/j.ajogmf.2021.100375. Epub 2021 Apr 20. PMID 33852969

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective observational study of 48 patients at Montefiore Medical Center. Recruitment commenced following IRB approval in FEB 2017 (first patient was enrolled July 1, 2017). Study recruitment was paused due to COVID from March 2020 to June 2020 and resumed from June 2020 to May 2021.
Pre-assignment Details: All 48 participants who enrolled were simultaneously monitored with the EUM Device and the typical tocodynamometer.
Groups:
- Pregnant Women: Pregnant women with singleton pregnancy with gestational age greater than or equal to 24 weeks were monitored simultaneously with two different devices to measure contractions: the EUM300 (electrical uterine myography) and tocodynamometry
Period: Overall Study
Arm/Group | Pregnant Women
Started | 48
Completed | 48
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pregnant Women: Pregnant women with singleton pregnancy with gestational age greater than or equal to 24 weeks.
  The EUM300 (electrical uterine myography): External monitor intended for the evaluation of electrical signals originating in the uterus, thus providing a tool for measuring uterine activity as well as fetal heart rate.
Arm/Group | Pregnant Women
Number analyzed (Participants) | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.17 (5.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 22
  White | 0
  More than one race | 0
  Unknown or Not Reported | 26
Region of Enrollment [Number; unit: participants]
  United States | 48

OUTCOME MEASURES:

1. Primary Outcome: Continuity in Readings of Contractions
Description: Continuity in readings of contractions, as measured in the number of minutes without a readable tracing in a sample tracing, between the novel EUM device and the external tocodynamometer (standard care) were assessed in pregnant preterm patients. An uninterpretable tracing was defined as any contraction, or any period of contractions, with unclear/uninterpretable baseline, peak onset/timing, height/peak, or duration of contraction.
Time Frame: within 4 hours of device application
Measure: Mean (Standard Deviation); unit: Number of minutes
Groups:
- EUM Device: Contractions monitored using the EUM device
- Tocodynamometer: Contractions monitored with tocodynamometer
Arm/Group | EUM Device | Tocodynamometer
Number analyzed (Participants) | 48 | 48
Number of minutes | 0 (0) | 0 (0)
Statistical Analysis 1: Comparison: EUM Device vs Tocodynamometer; Test type: Superiority; p = 0.75, t-test, 2 sided; Relative Rate = 0.95, 95% CI 2-sided [0.69 to 1.31]

2. Primary Outcome: Continuity in Readings of Fetal Heart Rate
Description: Continuity in Fetal Heart rate readings, as measured by the number of minutes without a readable tracing in a sample tracing between the novel EUM/EMG device and the external tocodynamometer (standard care) will be assessed in pregnant preterm patients. An uninterpretable tracing is defined as any period of fetal heart rate tracing with unclear/uninterpretable baseline, variability, onset/timing, peak, frequency, or duration of accelerations/decelerations
Time Frame: within 4 hours of device application
Population: Fetal Heart Rate data was not collected and therefore not analyzed
Arm/Group | EUM Device | Tocodynamometer
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Duration of labor evaluation, up to 15 weeks
Groups:
- Pregnant Women: pregnant women with gestational age 24-36 weeks and 6 days presenting with preterm contractions or induction or augmentation of preterm labor
Arm/Group | Pregnant Women
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 0/48
Other Adverse Events (participants affected / at risk) | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT02993354/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/54/NCT02993354/ICF_001.pdf